CLINICAL TRIAL: NCT02208414
Title: A Randomized Double-Blind Placebo-Controlled Crab Allergy Reduction Study Using Nambudripad Allergy Elimination Techniques in NTU Campus
Brief Title: Randomized Double-Blind Placebo-Controlled Crab or Shrimp Allergy Reduction Study Using Nambudripad Allergy Elimination Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201111069RID
Record Dates: First submitted 2013-01-02; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Food Allergies
Keywords: Food Allergies
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crab or shrimp (Experimental): Intervention: treated with crab and shrimp energy signature vial using NAET
  Interventions: Procedure: NAET
- Placebo (Placebo Comparator): Treated with water vial
  Interventions: Procedure: NAET

INTERVENTIONS:
Procedure: NAET — NAET with acupressure and/or chiropractic procedures with the participant holding crab and shrimp energy signature vial
  Arms: Crab or shrimp
Procedure: NAET — NAET with acupressure and/or chiropractic procedures with the participant holding water vial
  Arms: Placebo

SUMMARY:
Purpose of this study is to determine whether NAET procedures are effective in the treatment of crab or shrimp allergy.

Hypothesis: experimental group will show a significant improvement over the control group in allergic symptom, serum crab- or shrimp-specific IgE and skin test for crab or shrimp extract.

DETAILED DESCRIPTION:
Nambudripad allergy elimination techniques (NAET) were developed by Dr. Devi Nambudripad in 1983. Many patients have been relieved of allergy and allergy-related disease by this treatment.

Lack of well-controlled clinical study prevents NAET from being accepted as a treatment option in current medical system.

The aim of this project is to conduct a double blind-placebo controlled study of applying NAET to treat crab or shrimp allergy.

The parameters to be measured are allergic symptom, crab- or shrimp-specific IgE and skin test before and after NAET treatment

ELIGIBILITY:
Inclusion Criteria:

* Older or equal to 20 years old
* History of allergic to crab or shrimp
* Positive serum crab- or shrimp-specific IgE

Exclusion Criteria:

* History of anaphylactic shock
* On medication of anti-histamine or steroid
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in allergic symptoms at 6 months | before NAET and 6 months after NAET
  Symptoms when exposed to crab or shrimp which include symptoms of skin, eye, respiratory tract, gastrointestinal tract, cardiovascular system and others. The participants give score subjectively from 0 to 10 according to the severity of the symptoms.

SECONDARY OUTCOMES:
Serum crab- or shrimp-specific IgE | before NAET, 1 month, 3 months and 6 months after NAET
Skin test | before NAET, 1 month and 6 months after NAET
  Skin test for crab or shrimp extract

CONTACTS AND LOCATIONS:
Overall Officials: Cha Ze Lee, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan